CLINICAL TRIAL: NCT03318367
Title: A Pilot Study to Determine if the Use of a Virtual Reality Education Module Reduces Anxiety and Increases Comprehension in Patients Receiving Radiation Therapy
Brief Title: Virtual Reality Education Module in Reducing Anxiety and Increasing Knowledge in Patients With Prostate Cancer Undergoing Radiation Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study expired at the IRB
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 14D.354; JT 6320 (Other: JeffTrial Number)
Record Dates: First submitted 2017-06-22; First posted 2017-10-23 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Prostate
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (virtual reality education module) (Experimental): After undergoing a previously planned CT simulation scan, patients complete a virtual reality education module to learn more about radiation therapy for prostate cancer. Patients also complete questionnaires before and after the module.
  Interventions: Other: Educational Intervention

INTERVENTIONS:
Other: Educational Intervention — Complete virtual reality education module

SUMMARY:
This pilot clinical trial studies a virtual reality education module in reducing anxiety and increasing knowledge in patients with prostate cancer undergoing radiation therapy. A virtual reality education module may be useful in helping patients understand what they can expect to happen during their radiation treatments and help reduce stress relating to the radiation treatments.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if a virtual reality education module for prostate cancer patients is effective in increasing patient comprehension and decreasing patient anxiety related to radiation treatments.

SECONDARY OBJECTIVES:

I. This pilot study could have implications for a broader patient base undergoing radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* English speaking males capable of giving informed consent
* Must be able to read English language
* Receiving pre-treatment cone beam and volumetric modulated arc therapy (VMAT) for prostate cancer on the "A" or "B" treatment machines at the Bodine Center
* Must be able to walk two city blocks
* Must not have any auditory or visual deficits

Exclusion Criteria:

* If inclusion criteria are not met
* Previous radiation therapy treatment
* Employment in radiation oncology

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-08-06 (Actual); Primary Completion 2016-06-03 (Actual); Study Completion 2016-08-11 (Actual)

PRIMARY OUTCOMES:
Standard deviation for difference in questionnaire response from pre-education to post-education | Through study completion, an average of 2 years
  A one-sided one-sample t-test will be used to analyze the average change score (pre - post) for each questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Den, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Sidney Kimmel Cancer Center — http://www.kimmelcancercenter.org
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/